CLINICAL TRIAL: NCT05453929
Title: Effect of the Deep Neuromuscular Block on Postoperative Delirium in Elderly Patients Undergoing Lumbar Surgery
Brief Title: Deep Neuromuscular Block on Postoperative Delirium in Lumbar Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Korea University Guro Hospital (Other)
Responsible Party: Principal Investigator, Seok Kyeong Oh, Assistant Professor, Korea University Guro Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 2021GR0301
Record Dates: First submitted 2022-07-08; First posted 2022-07-12 (Actual); Last update posted 2025-01-03 (Actual); Status verified 2025-01

CONDITIONS: Lumbar Spine Disease
MeSH Terms: conditions — Spinal Diseases | interventions — Rocuronium

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Deep NMB (Experimental): A TOF count of 0, and a PTC of 1 to 3 will be maintained, as close to 2 twitches as possible
  Interventions: Drug: Rocuronium for deep NMB
- Moderate NMB (Active Comparator): A TOF count of 1 to 3 will be maintained, as close to 2 twitches as possible
  Interventions: Drug: Rocuronium for moderate NMB

INTERVENTIONS:
Drug: Rocuronium for deep NMB — Deep neuromuscular blockade will be maintained using continuous infusion of rocuronium.
  Other Names: Deep NMB
  Arms: Deep NMB
Drug: Rocuronium for moderate NMB — Moderate neuromuscular blockade will be maintained using continuous infusion of rocuronium.
  Other Names: Moderate NMB
  Arms: Moderate NMB

SUMMARY:
The effect of deep neuromuscular blockade (NMB) during spine surgery reduced postoperative pain and bleeding in recent studies. Therefore by reducing these two factors, which were the contributing factors for postoperative delirium, deep NMB is expected to reduce the postoperative delirium. This study was designed to determine whether the deep NMB lowered the incidence of delirium after lumbar surgery.

ELIGIBILITY:
Inclusion Criteria:

* Aged 70 and more;
* Scheduled for an elective lumbar spine surgery;
* ASA physical status 1-3

Exclusion Criteria:

* Diagnosed neuromuscular disorder;
* Contraindications to the study drug, e. g. known allergy or hypersensitivity, hypotension, bradycardia, higher grade atrioventricular block;
* Patient with pre-existing cognitive impairment or dementia

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 230 (Actual)
Dates: Start 2021-09-16 (Actual); Primary Completion 2024-12-20 (Actual); Study Completion 2025-01-02 (Actual)

PRIMARY OUTCOMES:
Delirium by CAM-ICU | from just after surgery at the PACU to post-operative 5 days
  Occurrence of delirium assessed by CAM-ICU during the post-operative 5 days

SECONDARY OUTCOMES:
Intramuscular pressure | intraoperative
  Intramuscular pressure at the para-spinal muscles
Peak inspiratory airway pressure | intraoperative
  Peak inspiratory airway pressure (mmHg)

CONTACTS AND LOCATIONS:
Overall Officials: Seok Kyeong Oh, MD, PhD, Principal Investigator — Korea University Guro Hospital
Locations (1):
- Seok Kyeong Oh, Seoul, Gangnam-gu, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Morino T, Hino M, Yamaoka S, Misaki H, Ogata T, Imai H, Miura H. Risk Factors for Delirium after Spine Surgery: An Age-Matched Analysis. Asian Spine J. 2018 Aug;12(4):703-709. doi: 10.31616/asj.2018.12.4.703. Epub 2018 Jul 27. PMID 30060380
- [Result] Oh SK, Kwon WK, Park S, Ji SG, Kim JH, Park YK, Lee SY, Lim BG. Comparison of Operating Conditions, Postoperative Pain and Recovery, and Overall Satisfaction of Surgeons with Deep vs. No Neuromuscular Blockade for Spinal Surgery under General Anesthesia: A Prospective Randomized Controlled Trial. J Clin Med. 2019 Apr 12;8(4):498. doi: 10.3390/jcm8040498. PMID 31013693
- [Result] Kang WS, Oh CS, Rhee KY, Kang MH, Kim TH, Lee SH, Kim SH. Deep neuromuscular blockade during spinal surgery reduces intra-operative blood loss: A randomised clinical trial. Eur J Anaesthesiol. 2020 Mar;37(3):187-195. doi: 10.1097/EJA.0000000000001135. PMID 31860601
- [Result] Taylor H, McGregor AH, Medhi-Zadeh S, Richards S, Kahn N, Zadeh JA, Hughes SP. The impact of self-retaining retractors on the paraspinal muscles during posterior spinal surgery. Spine (Phila Pa 1976). 2002 Dec 15;27(24):2758-62. doi: 10.1097/00007632-200212150-00004. PMID 12486343